CLINICAL TRIAL: NCT00132457
Title: Use of Self-collected Vaginal Swabs as an Innovative Approach to Facilitate Testing for Repeat Chlamydia Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-4274; U36/CCU319276
Record Dates: First submitted 2005-08-18; First posted 2005-08-22 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2010-01

CONDITIONS: Chlamydia Infections
Keywords: Chlamydia; screening; Sexually transmitted disease
MeSH Terms: conditions — Chlamydia Infections; Sexually Transmitted Diseases

INTERVENTIONS:
Procedure: Self-collected vaginal swab for chlamydia testing

SUMMARY:
The purpose of this study is to determine if, among women who were treated for a prior chlamydial infection, home-based, self-collected vaginal swabs can increase rescreening for chlamydia in comparison with rescreening in the clinic. The study design is two randomized trials with enrollment at multiple family planning clinics and sexually transmitted disease (STD) clinics following a common protocol.

DETAILED DESCRIPTION:
The study consists of two complementary trials, denoted as Part A and Part B. In Part A, women/girls who had a positive test for chlamydia will be enrolled when they visit the study clinics for treatment. After written informed consent is obtained, women will be randomly assigned to the Clinic Group, in which they will be advised to return to the clinic for rescreening for chlamydia, or the Home Group, in which women will be asked to collect a vaginal swab at home and mail it to the study laboratory for chlamydia testing. In part B, women who were tested and empirically treated for a chlamydial infection will be called if their tests were positive. Enrollment will be offered over the phone after verbal consent. Rescreening will be scheduled 3 months after treatment of the initial infection for women in both trials.

ELIGIBILITY:
Inclusion Criteria:

* Women/girls with a lab-confirmed genital chlamydia infection

Exclusion Criteria:

* Women who are pregnant, or are trying to conceive in the following 3 months.
* Women who are planning to move in the following 3 months or currently living outside the study areas.
* Inability to understand spoken English adequately to assure informed consent and compliance with study procedures.
* Self-reported HIV infection; other serious illnesses or disability.
* Self-reported allergy to macrolide antibiotics such as azithromycin.
* Referrals from providers or clinics other than the STD or family planning clinics, unless women are re-tested at the STD clinics and test positive for chlamydia.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1830 (Estimated)
Dates: Start 2003-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Percent of women rescreened for chlamydia

CONTACTS AND LOCATIONS:
Overall Officials: Fujie Xu, Principal Investigator — Centers for Disease Control and Prevention
Locations (3):
- United States (3):
  - Louisiana State University (LSU) Health Sciences Center, New Orleans, Louisiana
  - The Mississippi State Department of Health, Bureau of STD/HIV, Jackson, Mississippi
  - Washington University, St Louis, Missouri

REFERENCES:
- [Derived] Xu F, Stoner BP, Taylor SN, Mena L, Tian LH, Papp J, Hutchins K, Martin DH, Markowitz LE. Use of home-obtained vaginal swabs to facilitate rescreening for Chlamydia trachomatis infections: two randomized controlled trials. Obstet Gynecol. 2011 Aug;118(2 Pt 1):231-239. doi: 10.1097/AOG.0b013e3182246a83. PMID 21775837